CLINICAL TRIAL: NCT07261254
Title: Advancing Health Equity Via Basic Income + Early Childhood Systems Integration: An RCT of the Baby Bonus Program
Brief Title: Integrating Systems and Basic Income: Improving Outcomes for Families of Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Health Plan of San Mateo (Unknown); The Fidelity Charitable Trust (Unknown); Silicon Valley Community Foundation (Other); San Mateo County Health (Unknown); First 5 San Mateo County (Unknown); The Jackie Speier Foundation (Unknown); Valhalla Foundation (Other)
Responsible Party: Principal Investigator, Ryan Christopher Padrez, Clinical Associate Professor, Pediatrics - General, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 78517
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Income; Infant, Newborn; Mothers; Poverty; United States; Healthcare Disparities; Child Care; Child Health; Community Health Workers; Hispanic or Latino; Medicaid; Child Development; Social Services Utilization; Health Services Utilization
Keywords: Guaranteed Basic Income; Community Health Workers; Medicaid; Medi-Cal; Community Partners; Coordinated Care; Coordinated Services; randomized trial; surveys; infant, newborn; newborn nursery
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Coordinated Care (Experimental): Participants will receive coordinated Services via a Community Health Worker for 3 years in a hybrid format.
  Interventions: Behavioral: Community Health Worker
- Group B: Coordinated Care + Monthly Income Support (Experimental): Participants will receive the same coordinated services as in group A in addition to guaranteed basic income for 36 months.
  Interventions: Behavioral: Community Health Worker + Guaranteed Basic Income
- Group C: Standard of care (No Intervention): Participants in this group and will receive no treatment or intervention.

INTERVENTIONS:
Behavioral: Community Health Worker — A Community Health Worker will assist participants in navigating the medical system and connecting the participants to community services during the first three years of their child's life.
  Arms: Group A: Coordinated Care
Behavioral: Community Health Worker + Guaranteed Basic Income — A Community Health Worker will assist participants in navigating the medical system and connecting the participants to community services during the first three years of their child's life. Participants will also receive a monthly unconditional cash gift for the first three years of their child's life.
  Arms: Group B: Coordinated Care + Monthly Income Support

SUMMARY:
Early childhood is a critical period, laying the foundation for future growth and deveopment. This foundational period has an outsized effect, impacting health, well-being and achievement across one's lifespan. The U.S. lacks a cohesive early childhood system to support families with young children ages 0-5. The goal of this randomized controlled trial(RCT) is to test if community-based support via community health workers(CHWs) improves social and health services utilization, and child development. Furthermore, the trial will examine if income support enhances the impact of a CHW integrated system. Participants are English and Spanish speaking families with healthy newborns. This RCT was designed based on family priorities, community capacity and needs in a collective impact model. This trial is anchored at a university based children's hospital and involves many partners: families, county health, county leadership, a leading early childhood non-profit organization, the county's Medicaid managed care organization.

ELIGIBILITY:
Inclusion Criteria:

Caregiver Eligibility Criteria

* 18 and Older
* Family plans to reside in San Mateo County
* Does not plan to move from the County in the next year
* Speaks English and/or Spanish
* Cared for in Postpartum Maternity unit

Child Eligibility Criteria

* Baby is being cared for in well newborn nursery
* Child is enrolled in Medicaid
* 36 weeks or older
* To be discharged home in the custody of the caregiver

Exclusion Criteria:

Caregiver Exclusion Criteria

* Will not consent to share data via Epic/Study
* Caregiver has significant cognitive impairment
* Caregiver under contact isolation

Child Exclusion Criteria

* Sibling already enrolled in the Baby Bonus Study
* Child has significant genetic disorder issues at birth
* Child is a multiple (not a singleton)

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change in attendance at well-child visits | 12, 24 and 36 months
  Dates of visits for primary care in Health Plan of San Mateo (HPSM, the county-based Medicaid Managed Care organization) claims data.
Change in attendance at maternal postpartum follow-up visits | 12 months
  Dates of visits for postpartum checks in HPSM claims data.
Change in pediatric Emergency Department visits | 12 months, 24 months and 36 months
  Number of visits to the pediatric Emergency Department as per the HPSM claims data.
Change in referrals to Child Protective Services | 12 months, 24 months and 36 months
  Number of referrals to Child Protective Services in San Mateo County Human Services Agency administrative data.
Change in utilization of the Women Infants and Children program (WIC) - survey parents | Baseline, year 1, year 2, year 3
  Research coordinators will complete a phone survey with parents regarding WIC usage
Change in utilization of the Women Infants and Children program (WIC) - administrative data | Baseline, 12 months, 24 months and 36 months
  Administrative data from San Mateo County Family Health Services Agency regarding WIC usage
Change in utilization of Supplemental Nutrition Assistance Program (SNAP) services - survey parents | Baseline, year 1, year 2, year 3
  Research coordinators will complete a phone survey with parents regarding SNAP usage
Change in utilization of SNAP services - administrative data | Baseline, 12 months, 24 months and 36 months
  Administrative data regarding SNAP obtained from San Mateo County Human Services Agency.
Change in food insecurity scale score as measured by U.S. Household Food Security Survey Module | Baseline, year 1, year 2, year 3
  Research coordinators will complete a phone survey with parents regarding the U.S. Household Food Security Survey Module: Six-Item Short Form
Change in financial well-being scale score | Baseline, year 1, year 2, year 3
  Research coordinators will complete a phone survey with parents regarding consumer Financial Protection Bureau's (CFPB) Financial Well-Being Scale (10 of 12 items)
Number of participants who will be able or unable to cover a $400 unexpected expense. | Baseline, year 1, year 2, year 3
  Research coordinators will complete a phone survey with parents regarding CFPB Financial Well-Being Scale
Change in child developmental trajectory | Approximately 18 to 22 months, and approximately 30 to 34 months.
  Study team will invite participants to clinical lab where a trained assessor will complete the Bayley-III Development Assessment for each child.

SECONDARY OUTCOMES:
Change in parent depression scale score as measured by Patient Health Questionnaire (PHQ-9) | Baseline, year 1, year 2, year 3
  Research coordinators will administer the PHQ-9 survey to parents to evaluate parent depression level.
Change in diagnoses for mental and behavioral health services for the parent - claims data | Administrative data at baseline, 12, 24 and 36 months
  Assessed through claims data from HPSM Diagnosis ICD-10 of MH/BH diagnoses and BH utilization by provider type
Change in referrals for mental and behavioral health services for the parent - administrative data Family Health Services (FHS) | Administrative data at baseline, 12, 24 and 36 months
  Assessed through FHS Administrative Data: Maternal mental health referrals, BHRS Admin Data: Enrollment in BHRS mental health services.
Change in referrals for mental and behavioral health services for the parent - administrative data from Behavioral health and Recovery Services (BHRS) | Administrative data at baseline, 12, 24 and 36 months
  Assessed through BHRS Admin Data: Enrollment in BHRS mental health services.
Change in parent stress level | Year 1, year 2, year 3
  Research coordinators will administer the Parental Stress Index (PSI) to parents to evaluate the birthing parent's stress level.
Change in the breastfeeding duration | Baseline, Year 1, year 2
  Research coordinators will survey participants about the number of months breastfeeding.
Number of parents applying to childcare | Year 1, year 2, year 3
  Research coordinators will survey parents if they applied for childcare for their child.
Number of parents applying to preschool | Year 3
  Research coordinators will survey parents if they applied for preschool for their child.
Change in the purchase pattern for the child at home. | Year 1, year 2, year 3
  Research coordinators will survey parents about purchasing books, clothes, diapers, and toys for their child.
Change in parental involvement with child | Year 1, year 2, year 3
  Research coordinators will survey parents asking if they increased or decreased parental engagement activities with their child such as singing, sharing stories, encouraging behavior and preventing challenging behavior, building up child's interest, reading, and engaging in verbal skills.
Change in protective factors scale score as measured by Protective Factors Survey, 2nd Edition (PFS-2). | Baseline, year 1, year 2, year 3
  Research coordinators will administer the PFS-2 to parents.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Padrez, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egan-Dailey S, Gennetian LA, Magnuson K, Duncan GJ, Yoshikawa H, Fox NA, Noble KG. Child-directed speech in a large sample of U.S. mothers with low income. Child Dev. 2024 Nov-Dec;95(6):2045-2061. doi: 10.1111/cdev.14139. Epub 2024 Jul 29. PMID 39073390
- [Background] Rhodes, E. (2024, December 5). Insights from OpenResearch on the 2021 Expanded Child Tax Credit. Open Research. https://www.openresearchlab.org/findings/ctc
- [Background] Reyes-Velarde, A. (2024, January 30). They're getting $1,000 a month for 3 years. How guaranteed income is changing lives in L.A. County. CalMatters. http://calmatters.org/california-divide/2024/01/guaranteed-income-program/
- [Background] De Andrade, L. H. A., Ylikännö, M., & Kangas, O. (2021). Increased Trust in the Finnish UBI Experiment - Is the Secret Universalism or Less Bureaucracy? Basic Income Studies, 17(1), 95-115. https://doi.org/10.1515/bis-2021-0004
- [Background] Sauval M, Duncan GJ, Gennetian LA, Magnuson KA, Fox NA, Noble KG, Yoshikawa H. Unconditional Cash Transfers and Maternal Employment: Evidence from the Baby's First Years Study. J Public Econ. 2024 Aug;236:105159. doi: 10.1016/j.jpubeco.2024.105159. Epub 2024 Jul 5. PMID 40726482
- [Background] Rojas, N. M., Yoshikawa, H., Gennetian, L., Lemus Rangel, M., Melvin, S., Noble, K., Duncan, G., & Magunson, K. (2020). Exploring the experiences and dynamics of an unconditional cash transfer for low-income mothers: A mixed-methods study. Journal of Children and Poverty, 26(1), 64-84. https://doi.org/10.1080/10796126.2019.1704161
- [Background] Murray, M., Bridges, K., Solano, M., Greiner, K., & Woodward, J. (2023). Food RX + CHW: Investigating the Role of Community Health Workers to Close the Food Insecurity Gap. Annals of Family Medicine, 21(Suppl 1), 4231. https://doi.org/10.1370/afm.21.s1.4231
- [Background] Miller, S., Rhodes, E., Bartik, A., Broockman, D., Krause, P., & Vivalt, E. (2024). Does Income Affect Health? Evidence from a Randomized Controlled Trial of a Guaranteed Income (No. w32711; p. w32711). National Bureau of Economic Research. https://doi.org/10.3386/w32711
- [Background] Magnuson, K., Duncan, G., Yoshikawa, H., Yoo, P., Han, S., Gennetian, L. A., Fox, N., Halpern-Meekin, S., & Noble, K. (2024). Can Cash Transfers Improve Maternal Well-being and Family Processes among Families with Young Children? An Experimental Analysis. SSRN. https://doi.org/10.2139/ssrn.4955765
- [Background] Savage JS, Kling SMR, Cook A, Hess L, Lutcher S, Marini M, Mowery J, Hayward S, Hassink S, Hosterman JF, Paul IM, Seiler C, Bailey-Davis L. A patient-centered, coordinated care approach delivered by community and pediatric primary care providers to promote responsive parenting: pragmatic randomized clinical trial rationale and protocol. BMC Pediatr. 2018 Sep 4;18(1):293. doi: 10.1186/s12887-018-1263-z. PMID 30180831
- [Background] Yama CL, Rook JM. The Child Tax Credit-Tax Policy as Health Policy. JAMA Pediatr. 2024 Nov 1;178(11):1097-1098. doi: 10.1001/jamapediatrics.2024.3927. PMID 39348149
- [Background] Sircar NR, Friedman EA. Financial security and public health: How basic income & cash transfers can promote health. Glob Public Health. 2018 Dec;13(12):1878-1888. doi: 10.1080/17441692.2018.1460383. Epub 2018 Apr 6. PMID 29621932
- [Background] Siddiqi A, Rajaram A, Miller SP. Do cash transfer programmes yield better health in the first year of life? A systematic review linking low-income/middle-income and high-income contexts. Arch Dis Child. 2018 Oct;103(10):920-926. doi: 10.1136/archdischild-2017-314301. Epub 2018 Apr 28. PMID 29705725
- [Background] Noble KG, Magnuson K, Gennetian LA, Duncan GJ, Yoshikawa H, Fox NA, Halpern-Meekin S. Baby's First Years: Design of a Randomized Controlled Trial of Poverty Reduction in the United States. Pediatrics. 2021 Oct;148(4):e2020049702. doi: 10.1542/peds.2020-049702. Epub 2021 Sep 2. PMID 34475270
- [Background] Hart ER, Sperber JF, Troller-Renfree SV, Ortells-Faci P, Halpern-Meekin S, Sandre A, Noble KG. Mothers with low incomes view both individual and structural interventions as potentially helpful for supporting early child development. Sci Rep. 2024 Aug 7;14(1):18374. doi: 10.1038/s41598-024-68762-4. PMID 39112497
- [Background] Halpern-Meekin S, Gennetian LA, Hoiting J, Stilwell L, Meyer L. Monthly unconditional income supplements starting at birth: Experiences among mothers of young children with low incomes in the U.S. J Policy Anal Manage. 2024 Summer;43(3):871-898. doi: 10.1002/pam.22571. Epub 2024 Mar 2. PMID 39035030
- [Background] Gennetian LA, Duncan GJ, Fox NA, Halpern-Meekin S, Magnuson K, Noble KG, Yoshikawa H. Effects of a monthly unconditional cash transfer starting at birth on family investments among US families with low income. Nat Hum Behav. 2024 Aug;8(8):1514-1529. doi: 10.1038/s41562-024-01915-7. Epub 2024 Jun 21. PMID 38907028
- [Background] Das A, Osypuk TL, Yoo PY, Magnuson K, Gennetian LA, Noble KG, Bruckner TA. Poverty reduction and childhood opportunity moves: A randomized trial of cash transfers to low-income U.S. families with infants. Health Place. 2024 Sep;89:103320. doi: 10.1016/j.healthplace.2024.103320. Epub 2024 Aug 2. PMID 39096582
- [Background] Coker TR, Gregory EF, McCord M, Cholera R, Bakken H, Chapman S, Anwar E, Lee J, Henry S, Chamberlain LJ. Integrating community health workers in early childhood well-child care: a statement from the Pediatric Academic Societies Maternal Child Health: First 1,000 days Special Interest Group. BMC Prim Care. 2024 Sep 27;25(1):345. doi: 10.1186/s12875-024-02582-3. PMID 39333888
- [Background] Coker TR, Liljenquist K, Lowry SJ, Fiscella K, Weaver MR, Ortiz J, LaFontaine R, Silva J, Salaguinto T, Johnson G, Friesema L, Porras-Javier L, Guerra LJS, Szilagyi PG. Community Health Workers in Early Childhood Well-Child Care for Medicaid-Insured Children: A Randomized Clinical Trial. JAMA. 2023 May 23;329(20):1757-1767. doi: 10.1001/jama.2023.7197. PMID 37120800
- [Background] Agarwal SD, Cook BL, Liebman JB. Effect of Cash Benefits on Health Care Utilization and Health: A Randomized Study. JAMA. 2024 Nov 5;332(17):1455-1463. doi: 10.1001/jama.2024.13004. PMID 39037892
- See also: San Mateo County Baby Bonus Website — http://first5sanmateo.org/baby-bonus/